CLINICAL TRIAL: NCT01505088
Title: A Prospective, Multi-Center, Randomized, Double-Masked, Positive-Controlled Phase 3 Clinical Trial Designed to Evaluate the Safety and Efficacy of Iontophoretic Dexamethasone Phosphate Ophthalmic Solution Compared to Prednisolone Acetate Ophthalmic Suspension (1%) in Patients With Non-Infectious Anterior Segment Uveitis
Brief Title: Safety and Efficacy Study of Iontophoretic Dexamethasone Phosphate Ophthalmic Solution to Treat Non-Infectious Anterior Segment Uveitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGP-437-004
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Anterior Uveitis
Keywords: Iontophoresis; Non-Infectious Anterior Segment Uveitis; Ophthalmology
MeSH Terms: conditions — Uveitis, Anterior | interventions — prednisolone acetate; Ophthalmic Solutions; Sodium Chloride; Benzalkonium Compounds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iontophoretic Dexamethasone Phosphate Ophthalmic Solution (Experimental): Dexamethasone phosphate (40 mg/mL) solution delivered by iontophoresis treatment consisting of 4.0 mA-min at 1.5 mA on Day 0 and Day 7 with accompanying placebo eyedrops (saline solution) for up to 28 days.
  Interventions: Drug: 40 mg/mL Dexamethasone phosphate ophthalmic solution; Drug: Placebo Eyedrops
- Prednisolone Acetate Ophthalmic Suspension (1%) (Active Comparator): Placebo (100 mM sodium citrate buffer solution) iontophoresis treatment consisting of 4.0 mA-min at 1.5 mA on Day 0 and Day 7 with accompanying prednisolone acetate ophthalmic suspension (1%) (positive control) eyedrops for up to 28 days.
  Interventions: Drug: Prednisolone Acetate (1%) Eyedrops; Drug: 100 mM sodium citrate buffer solution

INTERVENTIONS:
Drug: 40 mg/mL Dexamethasone phosphate ophthalmic solution — Transscleral iontophoresis delivery of EGP-437 (dexamethasone phosphate formulated for ocular iontophoresis)
  Arms: Iontophoretic Dexamethasone Phosphate Ophthalmic Solution
Drug: Prednisolone Acetate (1%) Eyedrops — Prednisolone acetate (1%) eyedrops
  Arms: Prednisolone Acetate Ophthalmic Suspension (1%)
Drug: 100 mM sodium citrate buffer solution — Transscleral iontophoresis delivery of 100 mM Sodium citrate buffer solution
  Arms: Prednisolone Acetate Ophthalmic Suspension (1%)
Drug: Placebo Eyedrops — Placebo Eyedrops
  Other Names: Saline/ Benzalkonium Chloride (BAK) Ophthalmic Solution
  Arms: Iontophoretic Dexamethasone Phosphate Ophthalmic Solution

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ocular iontophoresis with dexamethasone phosphate ophthalmic solution EGP-437 using the EyeGate® II Drug Delivery System (EGDS) compared to prednisolone acetate ophthalmic suspension (1%) in patients with non-infectious anterior segment uveitis.

DETAILED DESCRIPTION:
Anterior uveitis is a disorder of the eye associated with intraocular inflammation of the anterior portion of the uvea, particularly the iris and/or ciliary body. It is distinct from other iterations of uveitis such as posterior, diffuse and intermediate uveitis although it is the most common form of uveitis and accounts for approximately 75% of cases.

In a Phase 1/2 study (EGP-437-001), the delivery of EGP-437 (40 mg/mL dexamethasone phosphate solution) at four different iontophoresis dose levels was studied in 40 subjects with non-infectious anterior segment uveitis. The study demonstrated that a single EGP-437 treatment: lowered anterior chamber cell (ACC) scores in the majority of patients without requiring additional treatment; produced low short-term systemic exposure to dexamethasone and dexamethasone phosphate; and produced the most beneficial effects in the 1.6 and 4.8 mA-min dose groups; and caused mainly minor AEs and no non-ocular systemic corticosteroid mediated effects were observed.

The Phase 3 study is intended to confirm and extend the results from the Phase 2 study. The study is designed to assess the safety and efficacy Ocular Iontophoresis with EGP-437 4.0 mA-min at 1.5 mA and accompanying placebo eyedrops in comparison to Ocular Iontophoresis with sodium citrate buffer solution 4.0 mA-min at 1.5 mA and accompanying prednisolone acetate (1%) eyedrops for the treatment of non-infectious anterior segment uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 12 to 85 years with a diagnosis of non-infectious anterior segment uveitis defined as an anterior chamber cell count of ≥ 11 cells
* Receive, understand, and sign a copy of the written informed consent form
* Be able to return for all study visits and willing to comply with all study-related instructions

Exclusion Criteria:

* Have uveitis of infectious etiology
* Have active intermediate or posterior uveitis
* Known positive HLA-B27 with a severe (4+) fibrinoid reaction
* Have previous anterior segment uveitis episode in the study eye ≤ 4 weeks prior to baseline visit
* Have used topical corticosteroid treatment in the study eye ≤ 48 hours prior to baseline visit
* Have used oral corticosteroid within the past 14 days prior to baseline
* Have received intravitreal or sub-Tenon corticosteroid treatment in the study eye within the past 6 months prior to baseline visit
* Currently using prescribed nonsteroidal anti-inflammatory agents (i.e., use of over-the-counter dosages is allowable) or prescribed immunosuppressive agents, unless the dose has been stable for the last six weeks and no change in dosing is anticipated for the duration of the study
* Have IOP ≥ 25 mmHg at baseline, a history of glaucoma, or require ocular anti-hypertensive medications in the study eye
* Be known steroid intraocular pressure responders in either eye
* Have open wounds/skin disease on the forehead area where the iontophoresis return electrode will be applied
* Have severe lesions of the eyelids or the ocular surface impeding the application of the iontophoresis applicator
* Have known allergy to dexamethasone or dexamethasone phosphate or any medication to be used in this study
* Have history or diagnosis of ocular herpes, corneal lesion of suspected herpetic origin, or Behçet's disease
* Have monocular or BCVA worse than 20/80 in the fellow eye
* Have optic neuritis of any origin
* Have clinically suspected or confirmed central nervous system or ocular lymphoma
* Planning to undergo elective ocular surgery during the study
* Have active hyphema, pars planitis, choroiditis, clinically significant macular edema, toxoplasmosis scar, or vitreous hemorrhage
* Have severe/serious ocular pathology or medical condition which may preclude study completion
* Have pacemaker and/or any other electrical sensitive support system
* Be pregnant or lactating female, or female of childbearing age and using inadequate birth control method
* Have participated in another investigational device or drug study within 30 days of baseline visit
* Have significant Fuch's Corneal Dystrophy

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with with ACC count of zero at Day 14 | At Day 14 (plus or minus two days) following the first study treatment
  Proportion of patients with ACC count of zero at Day 14

SECONDARY OUTCOMES:
Proportion of patients with ACC count of zero at Day 7 | At Day 7 (plus or minus two days) following the first study treatment
  Proportion of patients with ACC count of zero at Day 7
Proportion of patients with ACC count of zero at Day 28 | At Day 28 (plus or minus two days) following the first study treatment
  Proportion of patients with ACC count of zero at Day 28
Proportion of patients with ACC count of zero at Day 56 | At Day 56 (plus or minus seven days) following the first study treatment
  The proportion of patients with ACC count of zero at Day 56
Mean change from baseline in ACC count and score at Day 7 | At Day 7 (plus or minus two days) following the first study treatment
  Mean change from baseline in ACC count and score at Day 7
Mean change from baseline in ACC count and score at Day 14 | At Day 14 (plus or minus two days) following the first study treatment
  Mean change from baseline in ACC count and score at Day 14
Mean change from baseline in ACC count and score at Day 28 | At Day 28 (plus or minus two days) following the first study treatment
  Mean change from baseline in ACC count and score at Day 28
Mean change from baseline in ACC count and score at Day 56 | At Day 56 (plus or minus seven days) following the first study treatment
  Mean change from baseline in ACC count and score at Day 56
Proportion of subjects with ACC count and score reduction from baseline of one or more units at Day 7 | At Day 7 (plus or minus two days) following the first study treatment
  Proportion of subjects with ACC count and score reduction from baseline of one or more units at Day 7
Proportion of subjects with ACC count and score reduction from baseline of one or more units at Day 14 | At Day 14 (plus or minus two days) following the first study treatment
  Proportion of subjects with ACC count and score reduction from baseline of one or more units at Day 14
Proportion of subjects with ACC count and score reduction from baseline of one or more units at Day 28 | At Day 28 (plus or minus two days) following the first study treatment
  Proportion of subjects with ACC count and score reduction from baseline of one or more units at Day 28
Proportion of subjects with ACC count and score reduction from baseline of one or more units at Day 56 | At Day 56 (plus or minus seven days) following the first study treatment
  Proportion of subjects with ACC count and score reduction from baseline of one or more units at Day 56
Time to anterior chamber cell count and score of zero | Up to 56 days (plus or minus seven days) following the first study treatment
  Time to anterior chamber cell count and score of zero

CONTACTS AND LOCATIONS:
Overall Officials: John D. Sheppard, M.D., Principal Investigator — Virginia Eye Consultants
Locations (39):
- United States (39):
  - Department of Ophthalmology at University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Eye Center, Chandler, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Doheny Eye Medical Group, Los Angeles, California
  - Orange County Retina Medical Group, Santa Ana, California
  - Colorado Retina Associates, Golden, Colorado
  - Corneal Consultants of Colorado, Littleton, Colorado
  - Connecticut Retina Consultants, LLC, Bridgeport, Connecticut
  - Eye Center of Southern Connecticut, Hamden, Connecticut
  - Yale Eye Center, New Haven, Connecticut
  - The Eye Associates of Manatee, LLP, Bradenton, Florida
  - Levenson Eye Associates, Jacksonville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Logan Ophthalmic Research, Tamarac, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Advanced Eye Care, Fort Oglethorpe, Georgia
  - Illinois Retina Associates, Chicago, Illinois
  - Raj K. Maturi, M.D. PC, Indianapolis, Indiana
  - Ellsworth Uveitis and Retina Care, Ellsworth, Maine
  - Wilmer Eye Institute, Baltimore, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Massachusetts Eye Research and Surgery Institution, Cambridge, Massachusetts
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Tauber Eye Center, Kansas City, Missouri
  - Comprehensive Eye Care Ltd., Washington, Missouri
  - Metropolitan Eye Research and Surgery Institute, Palisades Park, New Jersey
  - The New York Eye and Ear Infirmary, New York, New York
  - Charlotte Eye Ear Nose and Throat Associates, Matthews, North Carolina
  - Casey Eye Institute, Portland, Oregon
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Mid-Atlantic Retina, Philadelphia, Pennsylvania
  - Southern College of Optometry, Memphis, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Houston Eye Associates, Houston, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Virginia Eye Consultants, Norfolk, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington